CLINICAL TRIAL: NCT04139655
Title: Colchicine Prevents Myocardial Injury After Non-Cardiac Surgery Pilot Study (COPMAN)
Brief Title: Colchicine Prevents Myocardial Injury After Non-Cardiac Surgery Pilot Study
Acronym: COPMAN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility
Sponsor: University of British Columbia (Other)
Collaborators: Providence Health & Services (Other); Vancouver Coastal Health (Other Government)
Responsible Party: Principal Investigator, Ron Ree, Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H19-02858
Record Dates: First submitted 2019-09-25; First posted 2019-10-25 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Myocardial Infarction; Myocardial Injury; Major Adverse Cardiac Events; Infectious Complications
Keywords: MINS; Colchicine; Myocardial Injury; Major Adverse Cardiac Events; Myocardial Injury after Non-Cardiac Surgery; MACE
MeSH Terms: conditions — Myocardial Infarction; Cardiovascular Diseases | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Randomized Control Pilot Study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine Group (Experimental): Administration of oral colchicine at 0.6 mg 1 hour prior to surgery, then 0.6 mg twice daily starting on the night after surgery for 7 days or until discharge from hospital, whichever occurs earlier. For patient under 60kg in body weight, daily dose will be 0.6 mg once daily. Medical and surgical management of the participant will be carried out under each institute's standard clinical practice.
  Interventions: Drug: Colchicine 0.6 mg
- Placebo Group (Placebo Comparator): Participants allocated to the control group will receive a placebo pill at the same dosing regimen as with treatment group. Perioperative and surgical care will not be different from standard clinical practice.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Colchicine 0.6 mg — Oral colchicine given at 0.6 mg 1 hour prior to surgery, then 0.6 mg twice daily starting on the night after surgery for 7 days or until discharge from hospital, whichever occurs earlier. For patient under 60kg in body weight, daily dose will be 0.6 mg once daily. Medical and surgical management of the participant will be carried out under each institute's standard clinical practice.
  Arms: Colchicine Group
Drug: Placebo oral tablet — Placebo oral tablet given at 0.6 mg 1 hour prior to surgery, then 0.6 mg twice daily starting on the night after surgery for 7 days or until discharge from hospital, whichever occurs earlier. For patient under 60kg in body weight, daily dose will be 0.6 mg once daily. Medical and surgical management of the participant will be carried out under each institute's standard clinical practice.
  Arms: Placebo Group

SUMMARY:
Perioperative Myocardial Infarction (PMI) is a major contributor to perioperative mortality and morbidity with overall incidence of 5-16%. It is associated with increased 30-day mortality of 11.6% vs 2.2% of patients without PMI in non-cardiac surgical patients. However, its recognition and diagnosis remains challenging as the typical symptoms and findings of ischemic MI may be masked by post-operative changes and pain management.

In this study, the investigators hope to determine if colchicine decreases the incidence of MINS in high risk surgical patients undergoing non-cardiac surgery and optimally establish colchicine as a viable therapy to improve perioperative cardiovascular outcome in those patients.

DETAILED DESCRIPTION:
Perioperative Myocardial Infarction (PMI) is a major contributor to perioperative mortality and morbidity with overall incidence of 5-16%. It is associated with increased 30-day mortality of 11.6% vs 2.2% of patients without PMI in non-cardiac surgical patients. However, its recognition and diagnosis remains challenging as the typical symptoms and findings of ischemic MI may be masked by post-operative changes and pain management.

To support early detection and diagnosis of myocardial injury in the perioperative setting, myocardial injury after non-cardiac surgery (MINS) has been recognized as an important prognostic marker independently associated with mortality and significant morbidity in the perioperative period. MINS is defined as prognostically relevant myocardial injury due to ischemia that occurs during or within 30 days after noncardiac surgery. Perioperative screening and monitoring of MINS is recommended by the most recent 2016 Canadian Cardiovascular Society (CCS) Guidelines. One study found of the MINS patients, only 41.8% of which filled universal definition of MI. This may suggest that screening for MINS in the Perioperative setting by detecting post-operative troponin rise is an important marker to prompt further investigation and closer monitoring.

However, despite efforts in recognition and establishment of MINS, there is still no consensus for the optimal management of MINS in addition to routine cardiac risk stratification. Common MI management options may be complicated by post-operative changes such as anemia, hypotension, hypoxemia, and use of routine anti-platelet and anticoagulation agents and invasive intervention is associated with high risk of complication and mortality in the perioperative period.

Colchicine is an alkaloid anti-inflammatory drug with well-established safety and adverse effect profile in various clinical settings including pericarditis and gout flare. Pharmacologically, colchicine inhibits beta-tubulin polymerization into microtubules, preventing activation and migration of neutrophils to achieve its anti-inflammatory effect. Clinically in the cardiac surgery patient population, colchicine has been shown in multiple meta-analyses to be efficacious in preventing post-operative atrial fibrillation, in treatment and prevention of pericarditis and post-pericardiotomy syndrome. In patients who are high risk for cardiovascular events, systemic review has shown reduction in cardiovascular mortality and myocardial infarction in some studies. Colchicine is an ideal agent in the perioperative period as it does not increase the risk of major bleeding, hepatic and renal toxicity, and there is only gastrointestinal discomfort at high doses.

In this study, the investigators hope to determine if colchicine decreases the incidence of MINS in high risk surgical patients undergoing non-cardiac surgery and optimally establish colchicine as a viable therapy to improve perioperative cardiovascular outcome in those patients.

Research Question: In the current clinical setting, is a larger, multi-centre randomised controlled trial comparing effect of perioperative oral colchicine administration versus placebo on incidence of MINS feasible?

This pilot study will inform many aspects of the future multi-centre trial. The pilot study will provide information on the recruitment rate of eligible patients and incidence of MINS on the recruited patient, which will allow the investigators to determine the sample size required in the large multi-centre trial to detect clinically relevant differences.

The pilot study will also provide information on the operational aspect of clinical trial, including initial patient enrolment and consent processes, data collection from electronic chart review. This will help refine the process and improve efficiency of the larger trial.

Lastly, information collected on side-effects of study drug (colchicine) would improve timely detection and treatment of the associated side effects (GI, myopathies, and blood dyscrasias), as well as expected drop-out rate from the larger trial due to intolerance of these side effects.

ELIGIBILITY:
Inclusion Criteria:

Any patient undergoing non-cardiac surgery is eligible if (s)he is:

* Aged 45 years of age or older
* Expected to be admitted for >48 hours
* Have a preoperative Brain natriuretic peptide (BNP) value of 92 or higher, or a N-terminal prohormone brain natriuretic peptide (NT-proBNP) value of 300 or higher,
* If a BNP or NT-proBNP is not available, then the patient must fulfill at least one of the criteria for moderate to high risk of perioperative myocardial injury (see below):

Moderate to high risk for perioperative myocardial injury criteria:

* History of coronary artery disease
* History of peripheral artery disease
* History of stroke
* Undergoing major vascular surgery
* Any 3 of the following 9 criteria:

  1. Age 70 years or greater
  2. Undergoing intraperitoneal, retroperitoneal, intrathoracic, or major orthopaedic surgery
  3. History of heart failure
  4. History of transient ischemic attack
  5. History of diabetes requiring insulin or oral hypoglycemic medications
  6. Hypertension
  7. Serum creatinine greater than 170 mmol/mL
  8. History of smoking within 2 years of surgery
  9. Undergoing urgent or emergent surgery

Exclusion Criteria:

Patients will be ineligible for the study if (s)he has:

* An allergy to colchicine
* Myelodysplastic syndrome
* An estimated glomerular filtration rate (eGFR) of less than 30 mL/min/1.73m2
* Anticipated post-operative administration of cyclosporine, ketoconazole, itraconazole, protease inhibitors, or clarithromycin

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Patients Recruited | 3 months
  The number of eligible subjects recruited in 3 months after 2 weeks of run-in period in participating centres

SECONDARY OUTCOMES:
Incidence of Myocardial Injury after Non-Cardiac Surgery (MINS) | From Post-Operatively day one up to 7 days post-operatively
  The incidence of MINS in the treatment versus placebo group, as defined by high sensitivity troponin T level > 65 ng/L or Troponin level > 0.03 ng/mL. The incidence of MINS will be determined upon review of the troponin assay on post-operative day 0, 1, 2 and 3rd (or according to each participating institution's own MINS pathway) and electrocardiogram (ECG) on post-operative day 1, or as otherwise clinically indicated and ordered by the perioperative team. Information will be obtained by review of blood work results and ECG on institution's electronic health record and patient's bedside chart if necessary by our research team member.
Adverse Events | Duration of hospital admission up to 7 days post-operatively
  We will collect adverse effects, whether or not associated with study drug through review of patient's bedside chart and discharge summary.
Incidence of premature discontinuation of the study drug and Reasoning | Post-Operatively until date of study drug discontinuation (up to 7 days post-operatively)
  Incidence of premature discontinuation of the study drug will be recorded. If the subject chooses to discontinue the study drug and withdraw from the study, the duration of treatment before withdraw as well as reasons of withdraw will be recorded.
Incidence of infectious complications | Duration of hospital admission up to 7 days post-operatively
  Incidence of infectious complications will also be recorded with review of chart and discharge summary. The determination of the complication will depend on patient's chart review, history and physical assessment by the primary care provider team, and associated imaging and laboratory investigations as clinically indicated. Complications include, but are not limited to: including but not limited to: pneumonia, surgical site infection, urinary tract infection, and sepsis during the hospital admission.

OTHER OUTCOMES:
Medical comorbidities | Duration of hospital admission up to 7 days post-operatively
  Based on patient charts.
Clinical risk stratification scores | Duration of hospital admission up to 7 days post-operatively
  Revised cardiac risk index (RCRI) scores based on patient charts. RCRI score is used and recommended by Canadian Cardiovascular Society as an evidence-based 30-day perioperative cardiovascular mortality and morbidity risk stratification tool. The tool is composed of 6 yes or no questions and provides a score from 0/6 to 6/6 which is interpreted as a percentage of 30-day risk of death, MI, or cardiac arrest. The lowest risk percentage is 3.9% and the highest percentage risk is 15%. A higher percentage indicates a higher risk of death, MI, or cardiac arrest in 30-days post-operatively.
Neutrophil to lymphocyte ratio (NLR) | Pre-operatively up to 7 days post-operatively
  Based on patient charts, to be obtained from patient's pre-operative bloodwork. NLR is a marker of neutrophil predominant inflammatory state that is associated with Major Adverse Cardiac Events (MACE) in a systemic review

CONTACTS AND LOCATIONS:
Overall Officials: Ron Ree, MD, Principal Investigator — Providence Health Care and UBC
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devereaux PJ, Xavier D, Pogue J, Guyatt G, Sigamani A, Garutti I, Leslie K, Rao-Melacini P, Chrolavicius S, Yang H, Macdonald C, Avezum A, Lanthier L, Hu W, Yusuf S; POISE (PeriOperative ISchemic Evaluation) Investigators. Characteristics and short-term prognosis of perioperative myocardial infarction in patients undergoing noncardiac surgery: a cohort study. Ann Intern Med. 2011 Apr 19;154(8):523-8. doi: 10.7326/0003-4819-154-8-201104190-00003. PMID 21502650
- [Background] Puelacher C, Lurati Buse G, Seeberger D, Sazgary L, Marbot S, Lampart A, Espinola J, Kindler C, Hammerer A, Seeberger E, Strebel I, Wildi K, Twerenbold R, du Fay de Lavallaz J, Steiner L, Gurke L, Breidthardt T, Rentsch K, Buser A, Gualandro DM, Osswald S, Mueller C; BASEL-PMI Investigators. Perioperative Myocardial Injury After Noncardiac Surgery: Incidence, Mortality, and Characterization. Circulation. 2018 Mar 20;137(12):1221-1232. doi: 10.1161/CIRCULATIONAHA.117.030114. Epub 2017 Dec 4. PMID 29203498
- [Background] Vascular Events In Noncardiac Surgery Patients Cohort Evaluation (VISION) Study Investigators; Devereaux PJ, Chan MT, Alonso-Coello P, Walsh M, Berwanger O, Villar JC, Wang CY, Garutti RI, Jacka MJ, Sigamani A, Srinathan S, Biccard BM, Chow CK, Abraham V, Tiboni M, Pettit S, Szczeklik W, Lurati Buse G, Botto F, Guyatt G, Heels-Ansdell D, Sessler DI, Thorlund K, Garg AX, Mrkobrada M, Thomas S, Rodseth RN, Pearse RM, Thabane L, McQueen MJ, VanHelder T, Bhandari M, Bosch J, Kurz A, Polanczyk C, Malaga G, Nagele P, Le Manach Y, Leuwer M, Yusuf S. Association between postoperative troponin levels and 30-day mortality among patients undergoing noncardiac surgery. JAMA. 2012 Jun 6;307(21):2295-304. doi: 10.1001/jama.2012.5502. PMID 22706835
- [Background] Botto F, Alonso-Coello P, Chan MT, Villar JC, Xavier D, Srinathan S, Guyatt G, Cruz P, Graham M, Wang CY, Berwanger O, Pearse RM, Biccard BM, Abraham V, Malaga G, Hillis GS, Rodseth RN, Cook D, Polanczyk CA, Szczeklik W, Sessler DI, Sheth T, Ackland GL, Leuwer M, Garg AX, Lemanach Y, Pettit S, Heels-Ansdell D, Luratibuse G, Walsh M, Sapsford R, Schunemann HJ, Kurz A, Thomas S, Mrkobrada M, Thabane L, Gerstein H, Paniagua P, Nagele P, Raina P, Yusuf S, Devereaux PJ, Devereaux PJ, Sessler DI, Walsh M, Guyatt G, McQueen MJ, Bhandari M, Cook D, Bosch J, Buckley N, Yusuf S, Chow CK, Hillis GS, Halliwell R, Li S, Lee VW, Mooney J, Polanczyk CA, Furtado MV, Berwanger O, Suzumura E, Santucci E, Leite K, Santo JA, Jardim CA, Cavalcanti AB, Guimaraes HP, Jacka MJ, Graham M, McAlister F, McMurtry S, Townsend D, Pannu N, Bagshaw S, Bessissow A, Bhandari M, Duceppe E, Eikelboom J, Ganame J, Hankinson J, Hill S, Jolly S, Lamy A, Ling E, Magloire P, Pare G, Reddy D, Szalay D, Tittley J, Weitz J, Whitlock R, Darvish-Kazim S, Debeer J, Kavsak P, Kearon C, Mizera R, O'Donnell M, McQueen M, Pinthus J, Ribas S, Simunovic M, Tandon V, Vanhelder T, Winemaker M, Gerstein H, McDonald S, O'Bryne P, Patel A, Paul J, Punthakee Z, Raymer K, Salehian O, Spencer F, Walter S, Worster A, Adili A, Clase C, Cook D, Crowther M, Douketis J, Gangji A, Jackson P, Lim W, Lovrics P, Mazzadi S, Orovan W, Rudkowski J, Soth M, Tiboni M, Acedillo R, Garg A, Hildebrand A, Lam N, Macneil D, Mrkobrada M, Roshanov PS, Srinathan SK, Ramsey C, John PS, Thorlacius L, Siddiqui FS, Grocott HP, McKay A, Lee TW, Amadeo R, Funk D, McDonald H, Zacharias J, Villar JC, Cortes OL, Chaparro MS, Vasquez S, Castaneda A, Ferreira S, Coriat P, Monneret D, Goarin JP, Esteve CI, Royer C, Daas G, Chan MT, Choi GY, Gin T, Lit LC, Xavier D, Sigamani A, Faruqui A, Dhanpal R, Almeida S, Cherian J, Furruqh S, Abraham V, Afzal L, George P, Mala S, Schunemann H, Muti P, Vizza E, Wang CY, Ong GS, Mansor M, Tan AS, Shariffuddin II, Vasanthan V, Hashim NH, Undok AW, Ki U, Lai HY, Ahmad WA, Razack AH, Malaga G, Valderrama-Victoria V, Loza-Herrera JD, De Los Angeles Lazo M, Rotta-Rotta A, Szczeklik W, Sokolowska B, Musial J, Gorka J, Iwaszczuk P, Kozka M, Chwala M, Raczek M, Mrowiecki T, Kaczmarek B, Biccard B, Cassimjee H, Gopalan D, Kisten T, Mugabi A, Naidoo P, Naidoo R, Rodseth R, Skinner D, Torborg A, Paniagua P, Urrutia G, Maestre ML, Santalo M, Gonzalez R, Font A, Martinez C, Pelaez X, De Antonio M, Villamor JM, Garcia JA, Ferre MJ, Popova E, Alonso-Coello P, Garutti I, Cruz P, Fernandez C, Palencia M, Diaz S, Del Castillo T, Varela A, de Miguel A, Munoz M, Pineiro P, Cusati G, Del Barrio M, Membrillo MJ, Orozco D, Reyes F, Sapsford RJ, Barth J, Scott J, Hall A, Howell S, Lobley M, Woods J, Howard S, Fletcher J, Dewhirst N, Williams C, Rushton A, Welters I, Leuwer M, Pearse R, Ackland G, Khan A, Niebrzegowska E, Benton S, Wragg A, Archbold A, Smith A, McAlees E, Ramballi C, Macdonald N, Januszewska M, Stephens R, Reyes A, Paredes LG, Sultan P, Cain D, Whittle J, Del Arroyo AG, Sessler DI, Kurz A, Sun Z, Finnegan PS, Egan C, Honar H, Shahinyan A, Panjasawatwong K, Fu AY, Wang S, Reineks E, Nagele P, Blood J, Kalin M, Gibson D, Wildes T; Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Writing Group, on behalf of The Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Investigators; Appendix 1. The Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Study Investigators Writing Group; Appendix 2. The Vascular events In noncardiac Surgery patIents cOhort evaluatioN Operations Committee; Vascular events In noncardiac Surgery patIents cOhort evaluatioN VISION Study Investigators. Myocardial injury after noncardiac surgery: a large, international, prospective cohort study establishing diagnostic criteria, characteristics, predictors, and 30-day outcomes. Anesthesiology. 2014 Mar;120(3):564-78. doi: 10.1097/ALN.0000000000000113. PMID 24534856
- [Background] Duceppe E, Parlow J, MacDonald P, Lyons K, McMullen M, Srinathan S, Graham M, Tandon V, Styles K, Bessissow A, Sessler DI, Bryson G, Devereaux PJ. Canadian Cardiovascular Society Guidelines on Perioperative Cardiac Risk Assessment and Management for Patients Who Undergo Noncardiac Surgery. Can J Cardiol. 2017 Jan;33(1):17-32. doi: 10.1016/j.cjca.2016.09.008. Epub 2016 Oct 4. PMID 27865641
- [Background] Parashar A, Agarwal S, Krishnaswamy A, Sud K, Poddar KL, Bassi M, Ellis S, Tuzcu EM, Menon V, Kapadia SR. Percutaneous Intervention for Myocardial Infarction After Noncardiac Surgery: Patient Characteristics and Outcomes. J Am Coll Cardiol. 2016 Jul 26;68(4):329-38. doi: 10.1016/j.jacc.2016.03.602. PMID 27443427
- [Background] Lennerz C, Barman M, Tantawy M, Sopher M, Whittaker P. Colchicine for primary prevention of atrial fibrillation after open-heart surgery: Systematic review and meta-analysis. Int J Cardiol. 2017 Dec 15;249:127-137. doi: 10.1016/j.ijcard.2017.08.039. Epub 2017 Sep 1. PMID 28918897
- [Background] Agarwal SK, Vallurupalli S, Uretsky BF, Hakeem A. Effectiveness of colchicine for the prevention of recurrent pericarditis and post-pericardiotomy syndrome: an updated meta-analysis of randomized clinical data. Eur Heart J Cardiovasc Pharmacother. 2015 Apr;1(2):117-25. doi: 10.1093/ehjcvp/pvv001. Epub 2015 Feb 19. PMID 27533981
- [Background] Papageorgiou N, Briasoulis A, Lazaros G, Imazio M, Tousoulis D. Colchicine for prevention and treatment of cardiac diseases: A meta-analysis. Cardiovasc Ther. 2017 Feb;35(1):10-18. doi: 10.1111/1755-5922.12226. PMID 27580061
- [Background] Hemkens LG, Ewald H, Gloy VL, Arpagaus A, Olu KK, Nidorf M, Glinz D, Nordmann AJ, Briel M. Cardiovascular effects and safety of long-term colchicine treatment: Cochrane review and meta-analysis. Heart. 2016 Apr;102(8):590-6. doi: 10.1136/heartjnl-2015-308542. Epub 2016 Feb 1. PMID 26830663